CLINICAL TRIAL: NCT04066608
Title: Cross-sectional Study on the Prevalence of Fatty Liver and Metabolic Risk Factors in an HIV-infected Population
Brief Title: Prevalence of Advanced Fibrosis in Patients Living With HIV
Acronym: FLASH
Status: Enrolling by invitation | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Jörn M. Schattenberg, Jörn Schattenberg, MD; Head of the Metabolic Liver Research Program, Johannes Gutenberg University Mainz
Other Study IDs: 18-00379
Record Dates: First submitted 2019-08-17; First posted 2019-08-26 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Fatty Liver Disease
Keywords: Non-invasive Diagnostics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Monocentric, cross-sectional study to define the prevalence of advanced fibrosis in an HIV infected outpatient population. Follow-up over 10 years to assess clinical relevance.

DETAILED DESCRIPTION:
Globally a shift in the spectrum of diseases has occurred. While in earlier year's infectious (communicable) disease were the main contributors to morbidity and mortality, today non-communicable diseases (NCD) exhibit a dramatic increase and have reached epidemic proportions, even in developing countries. Diabetes, cardiovascular disease, and cancer are the most frequent NCDs and the underlying risk factors including Insulin resistance, dyslipidemia and obesity have been increasing over the last decades. The current study explores the prevalence of advanced fibrosis in an HIV-infected outpatient study population.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age >18

Exclusion Criteria:

* pregnancy
* disease with expectation of life under 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient Study Population at the University Medical Center Mainz
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of significant hepatic fibrosis | 1 year
  Significant hepatic fibrosis defined as greater or equal to >8,2 kPa meassured by transient elastography using a Fibroscan

SECONDARY OUTCOMES:
Prevalence of hepatic steatosis | 1 year
  Hepatic steatosis defined as greater or equal to 275 db/m measured by controlled attenuation parameter (CAP) using a Fibroscan
Incidence of events of interest (clinical outcome) | 10 years
  Over the 10 year follow-up time, (1) overall mortality, (2) the incidence of AIDS-associated and defining diseases (according to the CDC classification) and (3) metabolic morbidity including incidence of cardiovascular disease (CVD), type 2 diabetes, hyperlipidemia, renal function impairment, arterial hypertension (according to the International Diabetes Federation Task Force on Epidemiology) and (4) liver related-morbidity (according to the EASL; https://easl.eu/wp-content/uploads/2018/10/Non-invasive-English-report.pdf)

OTHER OUTCOMES:
Quality of Life Meassures at Baseline and during Follow-up | 10 yeras
  Health-related quality of life will be measured and reported using generic (EQ-5D) and disease-specific tools (MOS-HIV)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center of the Johannes Gutenber Univeristy, Mainz
  - University Medical Center of the Johannes Gutenberg University, Mainz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] European Association for Study of Liver; Asociacion Latinoamericana para el Estudio del Higado. EASL-ALEH Clinical Practice Guidelines: Non-invasive tests for evaluation of liver disease severity and prognosis. J Hepatol. 2015 Jul;63(1):237-64. doi: 10.1016/j.jhep.2015.04.006. Epub 2015 Apr 21. No abstract available. PMID 25911335